CLINICAL TRIAL: NCT02992769
Title: A Nomogram to Predict the Risk of Axillary Metastases in Breast Cancer Patients With Axillary Ultrasound
Brief Title: Predict the Risk of Axillary Metastases in Breast Cancer Patients With Axillary Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Fengyan Yu, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: 201653
Record Dates: First submitted 2016-12-11; First posted 2016-12-14 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer Female
Keywords: Breast Cancer; Nomogram; Ultrasound; Axillary Metastases
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Axillary lymph node status is a vital prognostic factors in breast cancer patients and provides crucial information for making treatment decisions.This projective observational study is planned to identify risk factors for axillary metastases in breast cancer patients with axillary ultrasound and to construct a nomogram to predict the risk of axillary metastases in these patients.

DETAILED DESCRIPTION:
Breast carcinoma is the most common malignancy in women, accounting for 25% of all female cancer cases and 15% of all cancer-related deaths in the world.Lymph node metastasis is a multifactorial event. Among patients with a preoperative axillary ultrasound, almost 40% of patients are pathologically proved to be free from axillary metastasis.The purpose of this study is to develop a nomogram to evaluate the probability of axillary metastasis as a tool to support clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* female patients with primary breast cancer
* receiving a successful SLNB or ALND
* pathological diagnosed, without distant metastasis
* a clinically negative axilla

Exclusion Criteria:

* pregnancy
* neoadjuvant therapy
* previous ipsilateral axillary surgery
* inflammatory breast cancer

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 Years to 70 Years (Adult)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Axillary Metastases | 4 months to 1.5 year
  Surgical treatment for breast cancer patients include breast-conserving surgery or mastectomy with or without breast reconstruction. Intraoperative ALND is carried out when the SLNs are positive by intraoperative frozen section. Post-operative H&E permanent staining is administered to confirm the results of the frozen section. Serial H&E and immunohistochemistry stain (IHC) are only carried out when axillary metastases are not visible after H&E staining.

CONTACTS AND LOCATIONS:
Overall Officials: Fengyan Yu, M.D.,Ph.D, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun-Yat-Sen Memorial Hospital of Sun-Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Lyman GH, Temin S, Edge SB, Newman LA, Turner RR, Weaver DL, Benson AB 3rd, Bosserman LD, Burstein HJ, Cody H 3rd, Hayman J, Perkins CL, Podoloff DA, Giuliano AE; American Society of Clinical Oncology Clinical Practice. Sentinel lymph node biopsy for patients with early-stage breast cancer: American Society of Clinical Oncology clinical practice guideline update. J Clin Oncol. 2014 May 1;32(13):1365-83. doi: 10.1200/JCO.2013.54.1177. Epub 2014 Mar 24. PMID 24663048
- [Background] Bevilacqua JL, Kattan MW, Fey JV, Cody HS 3rd, Borgen PI, Van Zee KJ. Doctor, what are my chances of having a positive sentinel node? A validated nomogram for risk estimation. J Clin Oncol. 2007 Aug 20;25(24):3670-9. doi: 10.1200/JCO.2006.08.8013. Epub 2007 Jul 30. PMID 17664461
- [Background] Gentilini O, Veronesi U. Abandoning sentinel lymph node biopsy in early breast cancer? A new trial in progress at the European Institute of Oncology of Milan (SOUND: Sentinel node vs Observation after axillary UltraSouND). Breast. 2012 Oct;21(5):678-81. doi: 10.1016/j.breast.2012.06.013. Epub 2012 Jul 25. PMID 22835916
- [Background] Tucker NS, Cyr AE, Ademuyiwa FO, Tabchy A, George K, Sharma PK, Jin LX, Sanati S, Aft R, Gao F, Margenthaler JA, Gillanders WE. Axillary Ultrasound Accurately Excludes Clinically Significant Lymph Node Disease in Patients With Early Stage Breast Cancer. Ann Surg. 2016 Dec;264(6):1098-1102. doi: 10.1097/SLA.0000000000001549. PMID 26779976